CLINICAL TRIAL: NCT01928654
Title: Comparison Between Treatment With Yellow Micropulse Laser and Green Conventional Laser in Diabetic Macular Edema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luigi Sacco University Hospital (Other)
Responsible Party: Principal Investigator, Giovanni Staurenghi, MD, Luigi Sacco University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lasercomparison
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Diabetic Macular Edema
Keywords: Edema; Diabetic; Laser; Treatment
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micropulse laser treatment (Experimental): Sub-threshold laser treatment covering the area of retinal thickening with a dense pattern
  Interventions: Device: Micropulse laser treatment
- Laser modified ETDRS (Active Comparator): Macular treatment using the modified ETDRS protocol, with barely visible laser burns to close microaneurysms, or with a grid pattern in the area of retinal thickening.
  Interventions: Device: Laser modified ETDRS

INTERVENTIONS:
Device: Micropulse laser treatment — Device for subthreshold treatment of the retina, by decomposing a continuos wave of laser in micropulses, with 5% duty cycle, 200 milliseconds, 100 microns, and power adjusted according to patient's diopter transparency and pigmentation.
  Arms: Micropulse laser treatment
Device: Laser modified ETDRS — Device for visible treatment of the retina, with direct treatment of microaneurysms or grid pattern covering the area of retinal edema.
  Arms: Laser modified ETDRS

SUMMARY:
Macular edema is the most important cause of visual impairment in diabetic patients. Intravitreal injections of antiVEGF (vascular endothelial growth factor) agents and laser treatment are two effective therapies for stabilising visual acuity. However, antiVEGF therapy is very expensive and potentially needs to to be repeated for all patients life. Laser treatment, according to modified ETDRS (early treatment diabetic retinopathy study), produces retinal burns with possible negative consequences such as alterations in the visual fields.

With micropulse treatment modality laser energy is delivered in short pulses ("micropulses") rather than as a continuous wave. In this way the amount of energy delivered to the retina and retinal pigment epithelium (RPE) is significantly reduced. This finer control of the photothermal effects should avoid any retinal and RPE damage. At the same time, according to several published reports, the efficacy of treatment appears to be equivalent to conventional laser therapy.

Previous studies investigated the effects of 810nm micropulse laser therapy. Recently, this treatment modality has been made available also with 577nm wavelength, which corresponds to the maximum absorption level for blood. Aim of this study is to assess the safety and efficacy of 577nm micropulse laser treatment compared to conventional modified ETDRS laser therapy.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent prior to study entry
* male or female patients >= 18 years of age
* patients with diagnosis of diabetes type 1 or 2 and clinically significant macular edema
* visual impairment due to clinically significant diabetic macular edema
* best-corrected visual acuity included between 21 and 74 ETDRS letters
* central retinal thickness greater than 320 micron (Spectralis SD-OCT, Heidelberg Engineering, Germany)
* leakage and/or micro aneurysm in fluorescein angiography images within the area of retinal thickening
* HbA1C ≤10% with well-controlled blood pressure and renal function

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-10 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Mean change in visual acuity (ETDRS letters) | 12 months

SECONDARY OUTCOMES:
Mean change in central retinal thickness | 12 months
  Central retinal thickness corresponds to the mean retinal thickness within the 1-mm central subfield centred on the fovea. This measurement is obtained with Spectralis spectral-domain optical coherence tomography (SD-OCT) (Heidelberg Engineering, Germany).
Percentage of patients gaining ETDRS lines | 12 months
  Percentage of patients that gain 1, 2, or 3 ETDRS lines of visual acuity
Percentage of patients losing ETDRS lines | 12 months
  PErcentage of patients that loose 1, 2, or 3 ETDRS lines of visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Clinic - Luigi Sacco University Hospital, Milan, Italy